CLINICAL TRIAL: NCT05332275
Title: A Web-Based Media Parenting Intervention to Prevent Youth Substance Use
Brief Title: A Media Parenting Prevention Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB202301401; PRO00036387 (Other: University of Florida); IRB202101350 (Other: University of Florida); R34DA052793 (NIH)
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Substance Related Problem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - T.E.C.H. Parenting (Experimental): Intervention Arm participants will enroll in a web-based psychoeducational group (15 parents per group across 4 groups). Participants will receive psychoeducational information on media parenting, and they will be invited to participate in an online group discussion board to share their experiences with other parents in the intervention. In weeks 2-5, participants will learn about 4 domains of media parenting: 1) Talk to your child about media; 2) Educate your child about media-related risks; 3) Co-View/Co-Use media and technology actively with your child; and 4) establish House rules for media usage. Week 6 will review information and provide an "expert clinician" to support parent problem solving. Participants will receive 2-3 weekly push messages via text messaging prompting practice of skills learned in the group setting. Participants will be assessed at baseline, immediately following the 6 week intervention, and 3 months after the intervention is completed.
  Interventions: Behavioral: Intervention Arm - T.E.C.H. Parenting
- Control Arm - General Positive Parenting (Active Comparator): The Control Arm of the RCT is the attention control group. These participants will enroll in a web-based psychoeducational group (four groups of 15 parents each). They will receive 6 weeks of online psychoeducational material, including 2-3 push messages prompting skill practice. Parents will have access to an online discussion board to share experiences with other parents. This group will match the intervention arm of the study in number of study staff contacts, time of start/duration of the group, peer support, and availability of a professional in week six for consultation on parenting issues. Control participants will not receive information on media parenting. Participants in this group will be assessed at baseline, immediately following the six-week intervention period, and 3 months after intervention completion. Participants will be asked about exposure to TECH Parenting content at baseline and follow up to address potential contamination effects across study arms.
  Interventions: Behavioral: Control Arm - General Positive Parenting

INTERVENTIONS:
Behavioral: Intervention Arm - T.E.C.H. Parenting — Intervention Arm participants will enroll in a web-based psychoeducational group (15 parents per group across 4 groups). Participants will receive psychoeducational information on media parenting, and they will be invited to participate in an online group discussion board to share their experiences with other parents in the intervention. In weeks 2-5, participants will learn about 4 domains of media parenting: 1) Talk to your child about media; 2) Educate your child about media-related risks; 3) Co-View/Co-Use media and technology actively with your child; and 4) establish House rules for media usage. Week 6 will review information and provide an "expert clinician" to support parent problem solving. Participants will receive 2-3 weekly push messages via text messaging prompting practice of skills learned in the group setting. Participants will be assessed at baseline, immediately following the 6 week intervention, and 3 months after the intervention is completed.
  Arms: Intervention Arm - T.E.C.H. Parenting
Behavioral: Control Arm - General Positive Parenting — The Control Arm of the RCT is the attention control group. These participants will enroll in a web-based psychoeducational group (four groups of 15 parents each). They will receive 6 weeks of online psychoeducational material, including 2-3 push messages prompting skill practice. Parents will have access to an online discussion board to share experiences with other parents. This group will match the intervention arm of the study in number of study staff contacts, time of start/duration of the group, peer support, and availability of a professional in week six for consultation on parenting issues. Control participants will not receive information on media parenting. Participants in this group will be assessed at baseline, immediately following the six-week intervention period, and 3 months after intervention completion. Participants will be asked about exposure to TECH Parenting content at baseline and followup to address potential contamination effects across study arms.
  Arms: Control Arm - General Positive Parenting

SUMMARY:
Entertainment media commonly depict SU, and youth exposure to media SU is linked to youth initiation and progression of SU behavior. Parenting practices reduce exposure to and may mitigate risk associated with media depictions of SU, thus this research proposal will build upon current understanding of effective media parenting with the end goal of developing and testing a media parenting intervention designed to reduce youth risk for SU.

DETAILED DESCRIPTION:
Youth substance use (SU) is associated with many negative developmental outcomes including morbidity and mortality. Initiation of SU typically occurs during adolescence, and SU behavior often co-occurs with other risk behaviors (e.g., risky sexual behavior). Exposure to SU in the media is a well-documented influence on SU behavior, as it predicts early onset SU and progression to more problematic SU behavior. Media effects, while demonstrated to be consistent, stable, and strong even accounting for other social influences and personality characteristics, have received little attention in preventative SU research; yet youth exposure to media SU is a modifiable environmental risk for youth SU behavior. Parents can mitigate SU risk by limiting media SU exposures and intervening when youth are exposed. Parents report lack of media parenting skills, however, and no media parenting intervention designed specifically to reduce youth risk for SU exists. This project will examine the role of media parenting behaviors to reduce risk for early onset of youth SU. This program of research focuses on media depictions of SU, an important social and environmental influence implicated in the development, maintenance, and treatment of SU disorders. Specifically, the aims of this project are to target media-related mechanisms underlying SU initiation and associated risk factors as they relate to youth development. Improved understanding of specific parenting behaviors that contribute to prevention of youth SU, and mechanisms by which parenting behaviors may reduce risk related to media could inform the development of new and more effective interventions. Research aims in this application are designed to progress towards the end goal of developing a scalable, evidence-informed media parenting intervention to reduce youth risk for SU. The T.E.C.H. Parenting intervention will be tested in a sample of 120 parent participants (Aim 2 of grant protocol). Innovations include the use of web-based intervention content with supplemental push messaging to participants. Implementation data will be collected as part of the RCT to determine feasibility of web-delivered components of intervention content as well as usability and acceptability of intervention content from participants. This project is highly innovative in the use of technology to support parental engagement and dissemination of intervention. Further, web delivery of content provides an opportunity for parents to practice media parenting skills within the digital environment in a way that is adapted to the needs of the individual family and can be implemented in a range of diverse clinical settings.

ELIGIBILITY:
Inclusion Criteria:

Parents must

* have at least one middle school-aged child who resides with them
* be able to read at the 6th grade level in English
* have access to the internet and a smartphone to participate in web-based intervention groups and receive intervention push messages.

Exclusion Criteria:

-NA

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Media Parenting Behavior - Parent Report | Baseline up to Year 3
  The TECH Parenting measure is a 24 item indicator of general media parenting behaviors across four 6-item subscales: Talk; Educate; Co-Use; and House Rules. This measure has demonstrated reliability and predictive value for youth online risk behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Joy Gabrielli, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No